CLINICAL TRIAL: NCT05300685
Title: Peri-operative Oral Pain Control Following Buccal Graft Urethroplasty: Randomized Control Trial of Harvest Site Anesthetic
Brief Title: Peri-operative Oral Pain Control Following Buccal Graft Urethroplasty
Acronym: Buccal
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: MedStar Georgetown University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-35352
Record Dates: First submitted 2022-03-15; First posted 2022-03-29 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urethral Stricture, Male
Keywords: buccal urethroplasty; urethral stricture; urethroplasty; buccal block; lidocaine
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: This is a blinded, randomized, controlled trial following patients undergoing buccal urethroplasty (see criteria). This study will aim to assess three established anesthetic protocols for oral pain control. Each study arm holds equal weight.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Approximately 60 subjects will be randomized in a 1:1:1 ratio to receive 3 different local anesthetic regimens following buccal graft harvest. The care provider administering will not be masked to the type of block, but they will be blinded to the post op outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Standard of care (Active Comparator): 1. Prior to graft harvest - infiltration of 1% lidocaine with 1:100,000 epinephrine up to a maximum of 10 mL
  2. Routine, standard graft site hemostasis with monopolar cautery
  3. No suture closure of graft site
  4. No further infiltration of local anesthetic in mouth
  Interventions: Drug: Standard Buccal Harvest
- Group 2: Standard of care + Long acting local (Experimental): 1. Prior to graft harvest - infiltration of 1% lidocaine with 1:100,000 epinephrine up to a maximum of 10 mL
  2. Routine, standard graft site hemostasis with monopolar cautery
  3. No suture closure of graft site
  4. Up to a maximum of 10mL of 0.5% bupivacaine infiltration in the buccal graft site
  Interventions: Drug: Basic buccal procedure + Long acting local
- Group 3: Standard of care + Buccal block (Experimental): 1. Prior to graft harvest - infiltration of 1% lidocaine with 1:100,000 epinephrine up to a maximum of 10 mL
  2. Routine, standard graft site hemostasis with monopolar cautery
  3. No suture closure of graft site
  4. Up to a maximum of 10mL of 0.5% bupivacaine infiltration as a buccal block
  Interventions: Drug: Basic buccal procedure + Buccal block

INTERVENTIONS:
Drug: Standard Buccal Harvest — Our institutions current anesthetic regimen. Comparison group
  Arms: Group 1: Standard of care
Drug: Basic buccal procedure + Long acting local — Addition of long-acting local anesthetic to the wound bed following the oral graft harvest.
  Arms: Group 2: Standard of care + Long acting local
Drug: Basic buccal procedure + Buccal block — Addition of long-acting local anesthetic as a buccal block after oral graft harvest
  Arms: Group 3: Standard of care + Buccal block

SUMMARY:
Patients undergoing buccal urethroplasty will often have significant post-operative oral pain from the graft site. Various graft harvest techniques and methods for post-harvest hemostasis including graft site closure have been explored. Despite the frequency of this clinical scenario there is no established best practice for peri-operative pain management in this patient population. In addition to traditional post operative pain control, groups have sought various peri-operative anesthetic regimens to improve post operative pain. This has led recently to the description of various regional blocks including buccal and periorbital blocks for peri-operative local anesthetic. No study has looked at superiority of regional pain management in this patient population. This study will aim to assess three established anesthetic protocols for oral pain control in a blinded, randomized controlled trial.

Hypothesis: Patients who have buccal block will have lower post op pain without any increase adverse oral outcomes.

DETAILED DESCRIPTION:
This is a blinded, randomized, controlled trial following patients undergoing buccal urethroplasty (see criteria). This study will aim to assess three established anesthetic protocols for oral pain control. Each study arm holds equal weight. Approximately 60 subjects will be randomized in a 1:1:1 ratio to receive the following graft harvest techniques, which are all considered standard of care.

Group 1: Current Buccal Harvest

* Infiltration of lidocaine 1% with 1:100,000 epinephrine (maximum 10cc)
* Graft site hemostasis with monopolar cautery
* No suture closure of graft site

Group 2: Basic buccal procedure + Long acting local

* Infiltration of lidocaine 1% with epinephrine (maximum 10cc)
* Graft site hemostasis with monopolar cautery
* No suture closure of graft site
* 0.5% Marcaine (maximum 5cc) at case conclusion

Group 3: Basic buccal procedure + Buccal block

* Infiltration of lidocaine 1% with epinephrine (maximum 10cc)
* Graft site hemostasis with monopolar cautery
* No suture closure of graft site
* Buccal block with 0.5% Marcaine (maximum 5cc) at case conclusion

ELIGIBILITY:
Inclusion Criteria:

* Men, age 18 or older
* Undergoing anterior urethroplasty with buccal grafting
* Able to consent

Exclusion Criteria:

* Taking chronic opiates for pain
* Diagnosis of chronic pain
* Prior buccal urethroplasty
* Vulnerable population (e.g. prisoner)
* Renal dysfunction or allergy preventing NSAID use
* Liver dysfunction or allergy preventing Tylenol use
* Medical allergy to local anesthetic
* Medical allergy to Peridex/Magic Mouthwash
* NYHA Class III/IV
* Hematologic condition that excludes patient from surgery
* Post-operative complication resulting in inpatient stay
* Anesthetic complication
* No buccal site surgical complication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change(s) in Post-operative pain | Postoperative Day 1, 5, 10
  The Wong-Baker FACES pain scale is a validated scale where a score of 0 is no pain and 10 is the worst pain imaginable. Pain greater than or equal to 5 would result in significant limitations on daily life.
  Oral, incisional (surgical site), and overall pain will each be assigned a score of 0-10 at each time point (9 total scores).

SECONDARY OUTCOMES:
Change(s) in Post-operative Narcotic use | Postoperative Day 1, 5, 10
  Patient measure of number of oxycodone tablets taken (0-5). Patient request for additional narcotic medicaiton (Yes/No) Patient measure of adherence to non-narcotic pain regiman (Yes/No)

OTHER OUTCOMES:
Peri-operative Complications | Postoperative Day 0-30
  Clavien-Dingo is a validated tool to measure the severity of post-operative outcomes. Class I are mild and require no treatment. Class V is death.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Hampson, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - MedStar Urology, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonnavithula N, Bachu D, Sriramoju V, Devraj R, Gunta R, Pisapati MVLN. Effect of infraorbital nerve block on postoperative pain and 30-day morbidity at the donor site in buccal mucosal graft urethroplasty. J Anaesthesiol Clin Pharmacol. 2019 Jan-Mar;35(1):114-118. doi: 10.4103/joacp.JOACP_211_17. PMID 31057252
- [Background] Rourke K, McKinny S, St Martin B. Effect of wound closure on buccal mucosal graft harvest site morbidity: results of a randomized prospective trial. Urology. 2012 Feb;79(2):443-7. doi: 10.1016/j.urology.2011.08.073. Epub 2011 Nov 25. PMID 22119261
- [Background] Lumen N, Oosterlinck W, Hoebeke P. Urethral reconstruction using buccal mucosa or penile skin grafts: systematic review and meta-analysis. Urol Int. 2012;89(4):387-94. doi: 10.1159/000341138. Epub 2012 Aug 9. PMID 22889835

DOCUMENTS (1):
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT05300685/ICF_000.pdf